CLINICAL TRIAL: NCT02323022
Title: IAC Regimen Versus IA Regimen as Induction Treatment for Initially Diagnosed AML Patients: a Randomized Controlled Phase III Clinical Trial
Brief Title: Idarubicin Plus Cytarabine (IA) vs IA Plus Cladribine (IAC) as Induction Regimen to Treat Initially Diagnosed Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZ3202
Record Dates: First submitted 2014-12-12; First posted 2014-12-23 (Estimated); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IAC regimen (Experimental): Receive IAC induction therapy
  Interventions: Drug: IAC regimen
- IA regimen (Active Comparator): Receive an IA induction therapy
  Interventions: Drug: IA regimen

INTERVENTIONS:
Drug: IAC regimen — Induction treatment for initially diagnosed AML with IAC regimen, including Cladribine 5mg/msq/d (d1-5), Ara-C 100mg/msq/d(d1-7) and IDA 8mg/msq/d (d1-3)
  Arms: IAC regimen
Drug: IA regimen — Induction treatment for initially diagnosed AML with IAC regimen, including Ara-C 100mg/msq/d (d1-7) and IDA 12mg/msq/d (d1-3)
  Arms: IA regimen

SUMMARY:
The goal of this clinical trial is to compare the clinical efficacy and safety of IAC regimen and IA regimen as induction chemotherapy for initial diagnosed acute myeloid leukemia (AML) patients. The main question it aims to answer is:

•Does IAC regimen higher the complete remission rate in initial diagnosed AML patients? Researchers will compare IAC regimen to IA regimen to see if IAC works to treat AML.

Participants will:

* Receive IAC or IA as induction regimen
* Receive a second cycle of re-induction if partial remission
* Visit the clinic once every 3 to 6 months for assessment

ELIGIBILITY:
Inclusion Criteria:

* Initially diagnosed as AML (except APL)
* Aged between 18 and 60 year old
* Eastern Cooperative Oncology Group (ECOG) score no more than 3
* Informed consent file (ICF) signed

Exclusion Criteria:

* AML secondary to chronic leukemia and myeloproliferative neoplasms (MPNs)
* With other underlying malignancies
* Severe and uncontrolled infection
* Intolerant to the chemotherapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 618 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Complete Remission Rate | 1-2 months
  complete remission (CR) rate after the induction courses

SECONDARY OUTCOMES:
Overall Survival | 2 years
  2-year overall survival (OS)
Disease-Free Survival | 2 years
  2-year disease-free survival (DFS)
Cumulative Incidence of Relapse (CIR) | 2 years
  2-year cumulative incidence of relapse (CIR)

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, M.D., Ph.D., Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China